CLINICAL TRIAL: NCT05222490
Title: Collection of the Thermal Images of Diabetic Patients' Feet for FeetSee Device Performance Evaluation
Brief Title: FeetSee Thermal Images Collection Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetis JSC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RD-FS-01
Record Dates: First submitted 2021-11-25; First posted 2022-02-03 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Diabetic with Ulcers (Experimental): Patient with diabetic foot and ulceration diagnosed/confirmed by the study physician on the day of enrollment
  Interventions: Device: Thermal Camera images acquisition - FeetSee; Device: Thermal Camera images acquisition - Reference
- Diabetic without Ulcers (Experimental): Patient without ulcers diagnosed/confirmed by the study physician on the day of enrollment
  Interventions: Device: Thermal Camera images acquisition - FeetSee; Device: Thermal Camera images acquisition - Reference
- Control (Active Comparator): Generally Healthy Non-diabetic Subjects
  Interventions: Device: Thermal Camera images acquisition - FeetSee; Device: Thermal Camera images acquisition - Reference

INTERVENTIONS:
Device: Thermal Camera images acquisition - FeetSee — Thermal images will be collected according to the instructions for use of the Feetsee device.
Device: Thermal Camera images acquisition - Reference — After 15 minutes of resting, thermal images from the reference device will be collected according to their manufacturer

SUMMARY:
The purpose of this study is to collect thermal images of diabetic patients' feet to evaluate the performance of Feetsee - foot monitoring device for periodic evaluation of the temperature over the soles of the feet for signs of inflammation.

DETAILED DESCRIPTION:
The aim of this study is to collect a database of thermal images of the diabetic persons' feet, and non-diabetic control groups' feet images, which in turn will enable us to build a system based on a mobile thermal camera and a mobile application for possible indication of signs of inflammation in feet. Enrolled participants will undergo a detailed history and physical examination of the foot at the beginning of the procedure day. Then the thermal images of the patient's feet will be taken. Participants will be also asked to take thermal images of their feet according to very well-explained instructions provided by the sponsor. Thermal images using the reference thermal camera will be taken following the Feetsee thermal camera. The images will be unidentified, collected, and stored for the development and performance evaluation of the Feetsee device Algorithm. At the end of the study procedure, participants or their caregivers will receive a short questioner on their experience with using the study device.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

Group 1/2: Diabetic with/without ulcers

1. Male/Female, 18 years or older
2. Diagnosis of type 1 or type 2 Diabetes Mellitus, confirmed by a family physician or an endocrinologist.
3. Patient with or without history of previous foot ulcer, confirmed by a family physician or an endocrinologist
4. For Group 1: Patient with diabetic foot and ulceration diagnosed/confirmed by the study physician on the day of enrollment For Group 2: Patient without ulcers diagnosed/confirmed by the study physician on the day of enrollment
5. Must be able to read, understand and sign the Informed Consent Form Control: Generally Healthy Non-diabetic

1. Male/Female, 18 years or older 2. No diabetes mellitus or other diseases that may have signs of polyneuropathy or impaired blood circulation in the foot. 3.No damage to the skin or the soft tissues of the examined feet. 4. Must be able to read, understand and sign the Informed Consent Form

Exclusion Criteria:

1. Critical ischemia and/or deep ulceration (grades 4 or 5 according to Texas grading system).
2. Active Infection/Gangrene
3. Active malignancy
4. Immunosuppressive disease
5. History of alcohol or drug abuse
6. Pregnant women (verbal confirmation or confirmation obtained within current medical records)
7. Cognitive deficit
8. End-stage renal disease
9. History of amputation proximal to the Trans-metatarsal (TM) joint
10. Other issues that, at the discretion of the investigator, renders the subject ineligible for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Estimate of a difference in temperature between two feet per subject | through study completion, on average within of 1 year
  The primary outcome of this study is collecting of adequate thermal images from study groups' individuals using Feetsee device in order to develop and evaluate its performance to detect a temperature difference between two foot as a potential sign of inflammation and compare the camera performance to the reference camera.

SECONDARY OUTCOMES:
To evaluate the usability of FeeSee device by patient and healthcare providers | through study completion, an average of 1 year
  The evaluation of Feetsee device usability by patients or their healthcare providers using a a dedicated usability questioner.

CONTACTS AND LOCATIONS:
Locations (1):
- Inlita Santara CTC, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No